CLINICAL TRIAL: NCT02163941
Title: Meditation Training for Emotional Numbing in Post-traumatic Stress Disorder
Brief Title: Meditation for Emotional Numbing in Post-Traumatic Stress Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Brain & Behavior Research Foundation (Other); Mind and Life Institute, Hadley, Massachusetts (Other)
Responsible Party: Principal Investigator, Jennifer Mascaro, Instructor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00070643
Record Dates: First submitted 2014-06-11; First posted 2014-06-16 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Prolonged Post-traumatic Stress Disorder
Keywords: PTSD; empathy; meditation; compassion; inflammation; oxytocin; fMRI
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Compassion Training (Experimental): 8 weeks of training in Cognitively-Based Compassion Training (CBCT). Classes will meet once per week for 2 hours and participants will be asked to meditate at home for 20 minute each day.
  Interventions: Behavioral: Compassion Training

INTERVENTIONS:
Behavioral: Compassion Training
  Other Names: Cognitively-Based Compassion Training; CBCT

SUMMARY:
For individuals suffering from posttraumatic stress disorder (PTSD), the emotional numbing and isolation that are a core aspect of their suffering and consistently impedes remediation often remains after first-line treatments are administered. Few interventions have proven successful for enhancing the empathy and social connectedness that will ultimately allow patients to flourish, and the search for target therapies is made more difficult by the fact that very little is known about the underlying physiology of emotional numbing and social isolation. The proposed study is designed to (1) investigate the hormonal, neural and immunological biomarkers related to emotional numbing, and (2) test whether cognitively-based compassion training (CBCT), an intervention designed and proven to enhance empathy, will reduce emotional numbing and increase empathy and social connectedness in veterans. To this end, thirty medically healthy males diagnosed with PTSD who continue to report emotional numbing symptoms after prolonged exposure therapy will receive 8 weeks of training in CBCT. Prior to, and again after the training, the investigators will assess patients' levels of oxytocin, inflammation, and self-reported emotional numbing and social connectedness. The investigators will also assess their neural response during a video task that assesses their ability to accurately read others' emotions. The investigators hypothesize that oxytocin, neural activity, and inflammation will predict social numbing, isolation, and empathy, and also that CBCT will positively impact the social outcomes that will pave the way toward health and well-being.

DETAILED DESCRIPTION:
Thirty otherwise medically healthy males between the ages of 25 and 55 who have previously met criteria for PTSD and have undergone prolonged exposure therapy (PET) yet continue to report emotional numbing symptoms as a chief complaint will be assessed for baseline levels of plasma oxytocin (OT), markers of pro-inflammatory cytokines, total mRNA expression in peripheral blood mononuclear cells (PBMCs), self-reported emotional numbing and social connectedness, and empathy. Real-world social connectedness will be assessed using an Electronically Activated Recorder (EAR) for two days, which will randomly record 50 second snippets of audio every 9 minutes and which will allow for quantification of time spent with others. Measures of empathy will include empathic accuracy during a dynamic empathic accuracy (EA) video task, which asks participants to rate what story-tellers are feeling while they tell positively and negatively valenced autobiographical stories. Because previous studies have shown that PTSD may interfere with subtle social processing skills and because one of the primary aims of this proposal is to uncover specific biomarkers related to self-reported emotional numbing, the investigators will also assess eye gaze and arousal covariance (correlation between skin conductance of video subject and that of study participant) during the EA task. Following baseline assessments, participants will participate in 8 weeks of CBCT, which entails twice-weekly meetings consisting of didactic information sessions and approximately 20 minutes of CBCT practice. Participants will be asked to practice at home for 20 minutes per day, and will be given a audio compact discs to guide at-home meditation. Upon completion of CBCT (Time 2), and again after 8-12 weeks (Time 3), all Time 1 assessments will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* previously met criteria for PTSD
* completed front-line treatment such as prolonged exposure therapy
* continue to report emotional numbing symptoms as a chief complaint

Exclusion Criteria (at the discretion of the researchers):

* Self-reported psychotic symptoms, current major depression, or suicidal ideation
* Self-reported active alcohol or drug abuse within the past six months
* Self-reported depression serious enough to require hospitalization, or that resulted in a suicide attempt, within the last year.
* Self-reported auto-immune disease such as lupus, crohn's disease, irritable bowel syndrome, or rheumatoid arthritis.
* Self-reported use of psychotropic medication, including antidepressants, mood stabilizers, antipsychotics or chronic benzodiazepine therapy that has changed in the past 6 weeks.
* Self-reported use of any medication that might strongly affect your stress or immune systems, including non-steroidal anti-inflammatory agents, COX-2 inhibitors, corticosteroids, beta-blockers or statins.
* Claustrophobia
* Ferromagnetic implants contraindicated by functional MRI (fMRI) safety regulations

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Social connectedness | up to 3 months
  Self-report questionnaire assessment of social connectedness
Empathic Accuracy | up to 3 months
  objective performance assessing accuracy of reading others' emotions
Social Interactions | up to 3 months
  objective measures of time spent with others as measured by an audio sampling device

SECONDARY OUTCOMES:
messenger ribonucleic acid (mRNA) | up to 3 months
  gene expression related to inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Mascaro, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Background] Mascaro JS, Rilling JK, Tenzin Negi L, Raison CL. Compassion meditation enhances empathic accuracy and related neural activity. Soc Cogn Affect Neurosci. 2013 Jan;8(1):48-55. doi: 10.1093/scan/nss095. Epub 2012 Sep 5. PMID 22956676
- [Background] Desbordes G, Negi LT, Pace TW, Wallace BA, Raison CL, Schwartz EL. Effects of mindful-attention and compassion meditation training on amygdala response to emotional stimuli in an ordinary, non-meditative state. Front Hum Neurosci. 2012 Nov 1;6:292. doi: 10.3389/fnhum.2012.00292. eCollection 2012. PMID 23125828
- [Background] Pace TW, Negi LT, Adame DD, Cole SP, Sivilli TI, Brown TD, Issa MJ, Raison CL. Effect of compassion meditation on neuroendocrine, innate immune and behavioral responses to psychosocial stress. Psychoneuroendocrinology. 2009 Jan;34(1):87-98. doi: 10.1016/j.psyneuen.2008.08.011. Epub 2008 Oct 4. PMID 18835662
- [Background] Pace TW, Negi LT, Sivilli TI, Issa MJ, Cole SP, Adame DD, Raison CL. Innate immune, neuroendocrine and behavioral responses to psychosocial stress do not predict subsequent compassion meditation practice time. Psychoneuroendocrinology. 2010 Feb;35(2):310-5. doi: 10.1016/j.psyneuen.2009.06.008. Epub 2009 Jul 16. PMID 19615827